CLINICAL TRIAL: NCT05221229
Title: Feasibility Study of GLP-1 Analogues for the Optimization of Outcomes in High BMI Patients Undergoing AbLation for Atrial Fibrillation
Brief Title: Outcome of Overweight AF Patients Following Ablation With a Potential Weight Loss Medication ( GOAL-AF )
Acronym: GOAL-AF
Status: Active, not recruiting | Type: Observational
Sponsor: University Hospital Birmingham (Other)
Collaborators: University of Birmingham (Other)
Responsible Party: Principal Investigator, Manish Kalla, Consultant Cardiologist and Electrophysiologist, University Hospital Birmingham
Other Study IDs: RRK7604
Record Dates: First submitted 2021-12-17; First posted 2022-02-02 (Actual); Last update posted 2025-07-28 (Actual); Status verified 2025-07

CONDITIONS: Atrial Fibrillation; Recurrence; Overweight and Obesity; Liraglutide
Keywords: Atrial Fibrillation; Liraglutide; Ablation; Biomarkers; Heart MRI(CMR)
MeSH Terms: conditions — Atrial Fibrillation; Recurrence; Overweight; Obesity | interventions — Liraglutide; Referral and Consultation

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Blood samples will be taken from all patients as part of their routine care, including measurements for full blood count, urea and electrolytes, liver function test, and AF biomarkers panel.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Study Cohort: A total of 30 patients will be included in the study group after screening of inclusion and exclusion criteria. Patients will have upstream risk factors assessed at the clinic consultation and offered risk factor optimization advice. In addition, they will received daily Liraglutide injections for 13 weeks before and 52 weeks after ablation.
  Interventions: Drug: Liraglutide plus upstream risk factors modification advice and consultation

INTERVENTIONS:
Drug: Liraglutide plus upstream risk factors modification advice and consultation — Patients will be on treatment with daily injections of Liraglutide for a total of 65 weeks. During initial consultation for AF ablation, patients' BMI, risk factors status and baseline blood tests were performed and reviewed. Then the patients were discussed and encouraged to achieve optimal goal of risk factors modifications by non pharmacological and pharmacological measures.

SUMMARY:
Atrial Fibrillation (AF) is the most common abnormal heart rhythm(arrhythmia) affecting about one in 40 people in England. Patients with AF often have symptoms ranging from palpitations and breathlessness, and a small number of patients may develop heart failure. The major complication of AF is stroke, and this is effectively treated with blood thinning medications (anticoagulation).

AF symptoms can lead to significant decline in quality of life and can affect patients' ability to work and exercise. There are numerous treatments targeted at maintaining normal rhythm and preventing AF recurrence. These include medications and catheter ablation.

Ablation has been shown to be more effective than medications for the long-term control of AF, but its efficacy is significantly reduced by upstream conditions such as high blood pressure, obesity, diabetes, and poor fitness levels. This results in increased complications, repeat procedures, and increased AF recurrence or patients.

Research currently available has shown that intensive risk factor control with weight loss and increased fitness can reduce AF burden and improve results from ablation. However, achieving these targets outside of a clinical trial have been challenging. Recent data has shown that a new class of drug (Liraglutide) can result in significant weight loss over a 3-month period, and pre-treatment prior to liver transplant has improved results and patient recovery.

The overall aim of this study is to determine if accelerated weight loss by Liraglutide before AF ablation is feasible to base a future trial to inform if this approach improves outcomes and can be safely adopted into routine clinical practice.

DETAILED DESCRIPTION:
Patients meeting the inclusion criteria waiting for atrial fibrillation (AF) ablation in Queen Elizabeth Hospital of Birmingham will be invited for the study.

The investigators aim to recruit 30 patients who meet eligibility criteria. The study will be delivered by a dedicated research fellow, supported by a team of supervising clinical researchers. The research fellow will be responsible for recruitment, study data collection, and follow up. They will also be supported by clinical research nurses.

Timeline of the study for study participants:

At 1st visit (baseline): this visit will focus on collected baseline data (listed below), education on how to administer liraglutide (weight loss medication), and use the Kardia device

The following steps will be undertaken:

* Weight and height: this is standard of care
* Blood Tests: routine and additional blood tests will be taken for research
* Heart MRI: this is undertaken routinely in our clinical practice
* Provision of heart monitoring device(Kardia) and right atrial mapping will be performed: this is an additional step for the research study
* Patient reported outcome measures (PROMs) questionnaire will be completed: this is an additional step for the research study
* Liraglutide injection: the study participant will be trained to self administer this medication
* The baseline electrophysiological study (right atrial mapping) will be also be scheduled at this time point and will require an additional visit: this is a 30 minute procedure under sedation undertaken via a vein at the top of the right leg in the cardiac catheterisation laboratory (a recording of what takes place during this type of procedure will be available for patients to see before enrolment). This will be a day case procedure. The patient will not be able to drive for 48h after this procedure and will need to schedule 5-7 days off work.

At 2nd visit (13 weeks from baseline): this review time point will collect data after 13 weeks of treatment with Liraglutide

* Weight and height
* Blood Tests: these are extra blood tests done for research
* Heart MRI will be repeated: this is an extra test done for research and will require an extra visit to the hospital
* Then AF ablation with left mapping will performed as planned and right atrial mapping will be repeated at the time of AF ablation: this will be a planned admission separate to the visit for the heart MRI scan
* PROMs will be completed: this will not require an extra visit and will be done during the admission for the MRI or ablation

At 3rd visit (13 weeks from AF Ablation):

* Routine post ablation follow up in the outpatient clinic
* Remote review of Kardia recordings for AF recurrence will be performed.

At 4th visit (26 weeks from AF Ablation):

* This follow will be remote to avoid additional visits to the hospital
* Remote review of Kardia recordings for AF recurrence will be performed.

At 5th visit (39 weeks from AF Ablation):

* This follow will be remote to avoid additional visits to the hospital
* Remote review of Kardia recordings for AF recurrence will be performed.

At 6th visit (52 weeks from AF ablation): in person review and final follow up for the research study

* Weight and height check for BMI
* Review of Kardia ECG data
* PROM questionnaire for quality of life assessment
* All follow up after this will be as clinically indicated via the NHS clinic

Study design support

* The Birmingham Clinical Trials Unit has supported the design of this study with the primary outcome being feasibility of the treatment protocol
* We have also established an AF patient group with whom the study protocol, patient information sheet and consent forms have been reviewed, suggestions made and changes instituted.

ELIGIBILITY:
Inclusion criteria:

Patients with symptomatic paroxysmal or persistent Atrial Fibrillation on the waiting list for AF ablation at Queen Elizabeth Hospital Birmingham who

1. are more than 18 and less than 80 of age,
2. have paroxysmal or persistent AF,
3. symptomatic: palpitations, shortness of breath, feeling of an irregular pulse or pause in heart activity, light-headedness, or dizziness) despite pharmacological anti-arrhythmic agents (or inability to take medications) therefore making them eligible for ablation therapy,
4. are above BMI- 30 kg/m2

Exclusion criteria:

Any one of the followings;

1. unable to undergo CMR,
2. Patients who are currently treated with a weight losing drug - including Orlistat, GLP-1 analogues or have had/or awaiting bariatric surgery,
3. Type 1 diabetes,
4. Type 2 diabetes on DPP-IV inhibitor or insulin: as blood sugar will need close monitoring on GLP-1 and insulin,
5. Patients with decompensated liver disease, end-stage renal disease or eGFR <30, NYHA class III/IV heart failure or active malignancy,
6. Any malignancy within the last 2 years except skin malignancies,
7. Pregnancy,
8. Patients with a history of thyroid cancer or pancreatitis,
9. Patients with a needle phobia.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with Atrial Fibrillation and risk factors defined by eligibility criteria planning to go for AF ablation in Queen Elizabeth Hospital of Birmingham will be approached to enrol in our study.
Sampling Method: Probability Sample
Enrollment: 29 (Actual)
Dates: Start 2022-04-17 (Actual); Primary Completion 2025-06-30 (Actual); Study Completion 2026-06-01 (Estimated)

PRIMARY OUTCOMES:
Adherence to Liraglutide by AF patients before and after first-time ablation [Time Frame- 13 weeks before and 52 weeks after ablation] | 13 weeks before and 52 weeks after ablation
  Adherence to medication: will be measured by the proportion of patients who tolerate total cumulative dose of 657 mg and more of Liraglutide at the end of follow up period (minimal maintenance dose of 1.8mg over 365 days).
Number of participants recruited over recruitment period [Time Frame-39 weeks] | 39 weeks
  The internal audit data identified, over a 2-year period, 112 patients for first time ablation with a BMI above 30. There are no competing studies, and the investigators do not expect a recruitment period of more than 39 weeks.
Accelerated weight loss by Liraglutide on AF patients before first-time ablation and during one year follow-up [Time Frame- 13 weeks from recruitment and 52 weeks after ablation] | 13 weeks from recruitment and 52 weeks after ablation
  Weight loss: Body mass change will be measured using a single set of calibrated scales using a standardised protocol. Weight in kilograms will be measured to calculate Body Mass Index (BMI).
  The proportion of patients achieving >10% weight loss, 5-9% and < 5% weight loss will be calculated.

SECONDARY OUTCOMES:
Recurrence of AF after first-time AF ablation during one year follow-up [Time Frame- 52 weeks] | 52 weeks
  Time to first recurrence- any symptomatic or asymptomatic AF (>30s) beyond 12-weeks blanking post ablation as detected by Kardia recording
  Recurrence of AF will be defined as a heart rhythm with no discernible p waves and irregular RR intervals, when atrioventricular conduction is not impaired on a standard 12 lead ECG or a recording of a single lead ECG tracing of equal or more than 30 seconds, by Kardia recording.
AF burden after first-time AF ablation during one year follow-up [Time Frame-52 weeks] | 52 weeks
  AF burden will be quantified by twice daily and symptom-triggered (onset and termination) Kardia recordings which will be sent daily. The time of the recorded AF event will be taken as the onset of the episode, with the next recorded sinus rhythm taken as the offset. The duration of the all episodes will then be reported as percentage over predefined periods (13th-26th weeks, 27th-39th weeks, and 40th- 52nd weeks after ablation).
  AF burden will be reported as percentage of total observed time.
Changes in Epicardial Fat Volume as measured on heart MRI(CMR) [Time Frame- at baseline and 13 weeks] | Baseline and 13 weeks
  A standardised protocol is used for MRI acquisition of the heart. For the sequences, ECG triggering is used and patients are in a breath-hold for 10-12 seconds during the acquisition period. For a correct horizontal long axes of the heart in diastole, fast-spin T1-weighted sequences with oblique axial orientation are used to obtain cardiac adipose tissue scans. Images are also acquired in the short-axis view, which covers the heart from apex of the ventricles to the top of the atria. Area is quantified for each slice, and volume(cm^3) is calculated by multiplying each area by the thickness with no gap between images.
Changes in Left Atrial Fibrosis in percentage [Time Frame- at baseline and 13 weeks] | Baseline and 13 weeks
  A standardised protocol is used for MRI acquisition of the heart. For the sequences, ECG triggering is used and patients are in a breath-hold for 10-12 seconds during the acquisition period. For a correct horizontal long axes of the heart in diastole, fast-spin T1-weighted sequences with oblique axial orientation are used to obtain cardiac adipose tissue scans. Images are also acquired in the short-axis view, which covers the heart from apex of the ventricles to the top of the atria. Late Gadolinium Enhancement(15 min delayed images) will be acquired for final analysis. Then an open access rendering software, CEMRGAPP from King's College London, will be used to render images to produce left atrial fibrosis in percentage of left atrial volume.
Changes in AF biomarkers [Time Frame- at baseline and 13 weeks] | Baseline and 13 weeks
  For AF biomarkers, plasma will be used by taking additional EDTA tubes. Then they are to be spun down, components separated, frozen at -20 celsius at the hospital, then transferred to IBR building of Institute of Cardiovascular Science of University of Birmingham for ROCHE testing and long-term storage at -80 celsius. FGF-23(picograms/millilitres) and BMP-10(nanograms/millilitres) will be measured quantitatively according to ROCHE testing panel.
Adherence to Kardia Recording Requirements [Time Frame- 39 weeks] | 39 weeks
  Adherence to Kardia recording requirements: will be measured by calculating the percentage of patients who upload at least 2 recordings per day after 12 weeks blanking period following ablation up to the end of follow-up period.
Changes in electro-anatomic mapping data in right atrium [Time Frame -at baseline and 13 weeks] | Baseline and 13 weeks
  The electrical signals of the right atrium will be recorded in electrophysiology study at the baselline and at the time of ablation. These measurements will be analysed offline for specific markers of atrial fibrillation such as low voltage measured in millivolts and conduction velocity measured in centimeters per second.
Changes in patient reported outcome measures (AFEQT- AF Effect on QualiTy of life) [Time Frame- at baseline, 13 weeks from baseline and 52 weeks after ablation] | Baseline, 13 weeks from baseline and 52 weeks after ablation
  The effect of this treatment approach on quality of life will be measured by undertaking questionnaires at specific time points that have been designed and validated for patients with AF.

CONTACTS AND LOCATIONS:
Overall Officials: Manish Kalla, BSc, MBBS, MRCP, DPhil, Principal Investigator — University Hospital Birmingham NHS Foundation Trust
Locations (1):
- University Hospitals Birmingham NHS Foundation Trust, Birmingham, West Midlands, United Kingdom

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Win KZ, Armstrong M, Steeds RP, Kalla M. Feasibility study of Glucagon-like peptide-1 analogues for the optimization of Outcomes in obese patients undergoing AbLation for Atrial Fibrillation (GOAL-AF) protocol. Pilot Feasibility Stud. 2024 Feb 21;10(1):36. doi: 10.1186/s40814-024-01454-y. PMID 38383462